CLINICAL TRIAL: NCT02936154
Title: A Phase 1, Double Blind (Sponsor Open), Placebo-controlled, Multiple-dose Study To Evaluate The Tolerability, Safety And Pharmacokinetics Of A Modified Release Formulation Of Pf-06650833 Under Fed Condition In Healthy Adult Japanese Subjects
Brief Title: Study for MR Formulation of PF-06650833 in Healthy Adult Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: B7921006
Record Dates: First submitted 2016-08-08; First posted 2016-10-18 (Estimated); Last update posted 2018-10-05 (Actual); Status verified 2018-10

CONDITIONS: Healthy
MeSH Terms: interventions — 1-(((2S,3S,4S)-3-ethyl-4-fluoro-5-oxopyrrolidin-2-yl)methoxy)-7-methoxyisoquinoline-6-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 300 mg (Experimental)
  Interventions: Drug: PF-06650833
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PF-06650833
  Arms: 300 mg
Drug: placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the tolerability, safety and pharmacokinetics of PF-06650833 orally administered as modified release tablets in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy female subjects of non childbearing potential and/or male Japanese subjects between the ages of 20 and 55 years, inclusive.
2. Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).
3. Subject must have four Japanese grandparents who were born in Japan.
4. Evidence of a personally signed and dated informed consent document.
5. Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.
2. Any condition possibly affecting drug absorption (eg, gastrectomy).
3. A positive urine drug screen.
4. Smoking cigarettes with exceeding provided criteria.
5. History of regular alcohol consumption exceeding provided limitations.
6. Treatment with an investigational drug within a provided criteria.
7. Abnormal supine blood pressure.
8. Abnormal pulse rate.
9. Abnormal 12 lead ECG.
10. History of tuberculosis.
11. History of hepatitis or positive testing for HIV, hepatitis B surface antigen, hepatitis B surface antibodies, hepatitis B core antibodies, hepatitis C antibodies or syphilis.
12. Any medical history of disease (ie, Gilbert's disease).
13. Abnormal clinical laboratory test related to cardiac and skeletal muscle injury.
14. Male subjects with partners currently pregnant; unwilling or unable to use a highly effective method of contraception
15. Use of prescription or nonprescription drugs, vitaminic and dietary supplements within a specified duration.
16. Blood donation exceeding a provided limitation.
17. History of sensitivity to heparin or heparin induced thrombocytopenia.
18. History of cancer (other than treated basal cell and squamous cell carcinoma of the skin) in the previous 5 years.
19. Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
20. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
21. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing an AE/SAE | Day 18

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | Day 1 and Day 10
Area under the plasma concentration time curve for dosing interval (AUCtau) | Day 1 and Day 10
Time to peak concentration | Day 1 and Day 10
Clearance | Day 10
Volume of distribution | Day 10
Observed exposure accumulation ratio for AUCtau | Day 10
Observed exposure accumulation ratio for Cmax | Day 10
Minimum plasma concentration (Cmin) | Days 2, 4, 7 and 10
Fluctuation ratio (Cmax:Cmin) | Day 10
Mean residence time | Day 10
change from baseline in vital signs | Day 18
change form baseline in electrocardiogram (ECG) parameters | Day 18
Incidence of treatment emergent clinical laboratory abnormalities | Day 18

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- P-one Clinic, Keikokai Medical Corporation, Hachioji-shi, Tokyo, Japan

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7921006&StudyName=A+Phase+1%2C+Double+Blind+%28sponsor+Open%29%2C+Placebo-controlled%2C+Multiple-dose+Study+To+Evaluate+The+Tolerability%2C+Safety+And+Pharmacokinetics+Of+A+Modified+Release+Formulation+Of+Pf-06650833+Under+Fed+Condition+In+Healthy+Adult+Japanese+Subjects